CLINICAL TRIAL: NCT05657249
Title: Alternative Surveillance Program for Prospective Cohort of a Super-high Risk Group of Developing HCC
Brief Title: Alternative Surveillance Program for Patients With High Risk Group of HCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Severance Hospital (Other); The Catholic University of Korea (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jeong Hee Yoon, Clinical Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SNUH-2021-1084
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: US; MRI; HCC; surveillance; risk estimation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US & MRI (Experimental): All participants undergo biannual US (as a part of standard-of-care) and annual non-contrast focused MRI.
  Interventions: Diagnostic Test: Non-contrast focused MRI

INTERVENTIONS:
Diagnostic Test: Non-contrast focused MRI — non-contrast liver MRI focusing on HCC surveillance in a short scan time.
  Other Names: Focused MRI; Abbreviated MRI

SUMMARY:
In a high-risk group, ultrasonography at 6-month intervals and short-protocol magnetic resonance imaging at 1-year intervals were performed. sensitivity, specificity, positive and negative predictive values for very early stage HCC are compared between conventional (biannual US) and alternative surveillance test are compared

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis B or C
* Child-Pugh classification A
* HCC risk score >= -2.04
* have not diagnosed with HCC
* on surveillance program using US and negative on previous US within 6-8 months of enrollment
* sign informed consent

Exclusion Criteria:

* younger than 40 years or older than 70 years old
* history of HCC
* severe GFR or on HD/PD due to renal failure
* contra-indication of MRI
* congestive hepatopathy
* iron deposition
* pregnancy or nursing mother
* non-viral hepatitis or liver cirrhosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of alternative surveillance program (alternating focused MRI + US in 6 month interval) and conventional surveillance (biannual US) for HCC detection | up to one year
  per-patient sensitivity, specificity, positive predictive value, negative predictive value for very early stage HCC, early stage HCC, all stage of HCC/liver cancer.

SECONDARY OUTCOMES:
Comparison of annual focused MRI and biannual US for HCC detection | up to one year
  per-patient sensitivity, specificity, positive predictive value, negative predictive value for very early stage HCC, early stage HCC, all stage of HCC/liver cancer.
diagnostic yield for HCC | up to one year
  HCC incidence in the group and detection rate with either US or focused MRI
scan time of focused MRI | up to one month
  in room time, table time are manually recorded
comparison between false referral rates of biannual US and annual focused MRI | up to one year
  comparison between false positive report/finding for HCC in each surveillance modality.

OTHER OUTCOMES:
comparison between incidental findings between biannual US and annual focused MRI | up to one year
  comparison of incidental findings detected between biannual US and annual focused MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hee Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No